CLINICAL TRIAL: NCT05432284
Title: Behavioral Pharmacology of THC and Beta-Myrcene
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00329344; R01DA043475 (NIH)
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cannabis Use
MeSH Terms: interventions — Dronabinol; nabiximols; beta-myrcene

STUDY DESIGN:
Intervention Model Description: All participants will complete all dose conditions (study arms) in a randomized order
Who Masked: Participant, Outcomes Assessor
Masking Description: placebo controlled, double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Placebo (Placebo Comparator): Placebo (ambient air)
  Interventions: Drug: Placebo
- Vaporized high THC alone (Experimental): 30mg of vaporized pure THC
  Interventions: Drug: THC
- Vaporized low THC alone (Experimental): 15mg of vaporized pure THC
  Interventions: Drug: THC
- Vaporized low beta-myrcene (Experimental): 2mg of vaporized beta-myrcene
  Interventions: Drug: Beta-Myrcene
- Vaporized high beta-myrcene (Experimental): 9mg of vaporized beta-myrcene
  Interventions: Drug: Beta-Myrcene
- Vaporized low THC and low beta-myrcene (Experimental): 15mg vaporized THC with 2mg vaporized beta-myrcene
  Interventions: Drug: THC; Drug: Beta-Myrcene
- Vaporized low THC and high beta-myrcene (Experimental): 15mg vaporized THC with 9mg vaporized beta-myrcene
  Interventions: Drug: THC; Drug: Beta-Myrcene
- Vaporized high THC and low beta-myrcene (Experimental): 30mg vaporized THC with 2mg vaporized beta-myrcene
  Interventions: Drug: THC; Drug: Beta-Myrcene
- Vaporized high THC and high beta-myrcene (Experimental): 30mg vaporized THC with 9mg vaporized beta-myrcene
  Interventions: Drug: THC; Drug: Beta-Myrcene

INTERVENTIONS:
Drug: Placebo — Placebo (ambient air)
  Arms: Placebo
Drug: THC — Pure THC vapor
  Other Names: Cannabis
  Arms: Vaporized high THC alone; Vaporized high THC and high beta-myrcene; Vaporized high THC and low beta-myrcene; Vaporized low THC alone; Vaporized low THC and high beta-myrcene; Vaporized low THC and low beta-myrcene
Drug: Beta-Myrcene — Pure beta-myrcene vapor
  Arms: Vaporized high THC and high beta-myrcene; Vaporized high THC and low beta-myrcene; Vaporized high beta-myrcene; Vaporized low THC and high beta-myrcene; Vaporized low THC and low beta-myrcene; Vaporized low beta-myrcene

SUMMARY:
This study will evaluate the pharmacokinetics and pharmacodynamics of vaporized b-myrcene and THC administered via inhalation.

DETAILED DESCRIPTION:
The proposed study will be conducted at the Johns Hopkins Behavioral Pharmacology Research Unit (BPRU). Participants will complete 9 acute drug administration periods in which they will administer THC alone, myrcene alone, THC and myrcene together, or placebo. Subjective drug effects and vital signs will be assessed following drug administration. Each participant will receive all 9 dose conditions in a randomized order using a placebo controlled within-subject crossover design. The study will help us understand the individual and interactive effects of THC and b-myrcene, two common constituents found in cannabis.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be between the ages of 18 and 55
3. Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
4. Test negative for drugs of abuse other than cannabis, including breath alcohol at the screening visit and at clinic admission
5. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
6. Have a body mass index (BMI) in the range of 18 to 36 kg/m2
7. Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
8. Have no allergies to any of the ingredients used to prepare vapor (delta 9-THC, myrcene).
9. Demonstrate competency on cognitive performance measures at screening visit (e.g., PASAT score over 75).

Exclusion Criteria:

1. Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine 3 month prior to the Screening Visit;
2. History of or current evidence of significant medical (e.g. seizure disorder) or psychiatric illness (e.g. psychosis) judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
3. Use of an OTC, systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
4. Use of a prescription medication (with the exception of birth control prescriptions) within 5 half-lives for that specific drug; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
5. Cannabis use that is inconsistent with protocol requirements.
6. Clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
7. Individuals with anemia or who have donated blood in the prior 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Self-reported Drug Effect as assessed by the Drug Effect Questionnaire (DEQ) | 6 hours
  Peak rating (0-100) of Drug Effect on the DEQ, with 0 being no effect and 100 being maximum effect.

SECONDARY OUTCOMES:
Self-reported "Tired/Sleepy" as assessed by the Drug Effect Questionnaire (DEQ) | 6 hours
  Peak rating (0-100) of Tired/Sleepy on the DEQ, with 0 being no effect and 100

OTHER OUTCOMES:
Driving performance as assessed by composite drive score | .5 hours
  Driving impairment will be assessed via a composite drive score (higher scores indicate greater impairment). The composite drive score is derived by integrating various driving outcomes. There is no upper or lower limit to possible scores
Psychomotor performance as assessed by the Digit Symbol Substitution Task (DSST) | 6 hours
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Total correct trials in 90-seconds. Minimum score of 0 but no maximum score (higher scores indicate better performance).
Working memory performance as assessed by the Paced Auditory Serial Addition Task | 6 hours
  Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. Total correct trials out of 90 recorded is primary outcome (higher scores indicate better performance).
Heart rate | 6 hours
  Heart rate (beats/minute) will be measured while sitting down using the vitals machine.
Quantitative levels of D-9-THC in blood | 3 hours
  Blood is collected through an intravenous catheter, quantitative results are reported in nanograms per milliliter (ng/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No